CLINICAL TRIAL: NCT03679559
Title: Exercise to Improve Health and Quality-of-Life in Breast Cancer Survivors: A Feasibility Pilot Trial
Brief Title: Exercise in Improving Health and Quality of Life in Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: I 32816; NCI-2018-00455 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 32816 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2018-09-18; First posted 2018-09-20 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Invasive Breast Carcinoma
MeSH Terms: interventions — Practice Guidelines as Topic; Standard of Care; Resistance Training; Monitoring, Physiologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Arm I (home-based walking program, resistance training) (Experimental): Participants wear Fitbit, receive home-based DVD containing instructions to warm-up and cool-down, and brisk walk 30 minutes per day 5 days a week in order to achieve the 150 minutes per week of moderate intensity exercise. Participants also receive resistance training by watching the illustration video and completing 6 total blocks of 2-week per block exercise using the Thera-BandR exercise bands.
  Interventions: Behavioral: Exercise Intervention (home walking program and resistance training); Behavioral: Exercise Intervention (HIIT program and resistance training); Other: Informational Intervention; Other: Laboratory Biomarker Analysis; Device: Monitoring Device; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (home-based Zumba program, resistance training) (Experimental): Participants wear Fitbit and receive a XBOX system and the video game to strive for at least 3 50-minute medium or high intensity classes per week over 12 weeks. Participants may also take 20-minute classes or a mixture of 50- and 20-minute classes to meet the target. Participants receive resistance training as in Arm I.
  Interventions: Behavioral: Exercise Intervention (home-based Zumba program and resistance training); Other: Informational Intervention; Other: Laboratory Biomarker Analysis; Device: Monitoring Device; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm III (HIIT, resistance training) (Experimental): Participants wear Fitbit and attend supervised HIIT exercise sessions 3 days per week over 12 weeks. Participants receive resistance training as in Arm I.
  Interventions: Behavioral: Exercise Intervention (HIIT program and resistance training); Other: Informational Intervention; Device: Monitoring Device; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm IV (supervised moderate intensity walking program) (Active Comparator): Participants wear Fitbit and attend supervised moderate intensity walking sessions weekly for 50-60 each over 12 weeks. Participants undergo resistance training as in Arm I.
  Interventions: Behavioral: Exercise Intervention (HIIT program and resistance training)
- Arm V (usual physical activity) (Active Comparator): Participants wear Fitbit and continue their usual physical activity over 12 weeks.
  Interventions: Other: Best Practice

INTERVENTIONS:
Other: Best Practice — Continue usual physical activity
  Other Names: standard of care; standard therapy
  Arms: Arm V (usual physical activity)
Behavioral: Exercise Intervention (home walking program and resistance training) — Complete home-based walking program and resistance training
  Arms: Arm I (home-based walking program, resistance training)
Behavioral: Exercise Intervention (home-based Zumba program and resistance training) — Complete home-based Zumba program and resistance training
  Arms: Arm II (home-based Zumba program, resistance training)
Behavioral: Exercise Intervention (HIIT program and resistance training) — Complete HIIT program and resistance training
  Arms: Arm I (home-based walking program, resistance training); Arm III (HIIT, resistance training); Arm IV (supervised moderate intensity walking program)
Other: Informational Intervention — Watch video
  Arms: Arm I (home-based walking program, resistance training); Arm II (home-based Zumba program, resistance training); Arm III (HIIT, resistance training)
Other: Laboratory Biomarker Analysis — Correlative studies
  Arms: Arm I (home-based walking program, resistance training); Arm II (home-based Zumba program, resistance training)
Device: Monitoring Device — Wear Fitbit
  Other Names: Monitor
  Arms: Arm I (home-based walking program, resistance training); Arm II (home-based Zumba program, resistance training); Arm III (HIIT, resistance training)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
  Arms: Arm I (home-based walking program, resistance training); Arm II (home-based Zumba program, resistance training); Arm III (HIIT, resistance training)
Other: Questionnaire Administration — Ancillary studies
  Arms: Arm I (home-based walking program, resistance training); Arm II (home-based Zumba program, resistance training); Arm III (HIIT, resistance training)

SUMMARY:
This randomized pilot trial studies how well exercise works in improving health and quality of life in breast cancer survivors. Participating in an exercise program to maintain physical activity may help to improve health and quality of life in breast cancer survivors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the feasibility of conducting a 12-week preference option randomized exercise intervention program in breast cancer survivors.

SECONDARY OBJECTIVE:

I. To assess the adherence rate of each of the four 12-week intervention programs by breast cancer survivors in a randomized treatment arm and a patient preference arm.

OUTLINE: Participants are randomized into 1 of 5 arms.

ARM I: Participants wear Fitbit, receive home-based DVD containing instructions to warm-up and cool-down, and walk 10000 steps per day over 12 weeks in order to achieve the 150 minutes per week of moderate intensity exercise. Participants also undergo resistance training by watching the illustration video and completing 6 total blocks of 2-week per block exercise using the Thera-BandR exercise bands.

ARM II: Participants wear Fitbit and receive a XBOX system and the video game to strive for at least 3 50-minute medium or high intensity classes per week over 12 weeks. Participants may also take 20-minute classes or a mixture of 50- and 20-minute classes to meet the target. Participants undergo resistance training as in Arm I.

ARM III: Participants wear Fitbit and attend supervised High Intensity Interval Training (HIIT) exercise sessions 3 days per week over 12 weeks. Participants undergo resistance training as in Arm I.

ARM IV: Participants wear Fitbit and attend supervised moderate intensity walking sessions weekly for 50-60 each over 12 weeks. Participants undergo resistance training as in Arm I.

ARM V: Participants wear Fitbit and continue their usual physical activity over 12 weeks.

After completion of study intervention, participants are followed up at 2 weeks and 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure
* Have a previous history of invasive breast cancer who have completed treatment except for hormonal therapy and zoledronic acid (Zometa)
* Do not meet the United States (U.S.) Center for Disease Control and Prevention's physical activity guidelines (150 minutes or 2 hours and 30 minutes a week of moderate-intensity exercise)
* Meets criteria for participation in low to moderate risk exercise based on the American College of Sports Medicine guideline (ACSM)

Exclusion Criteria:

* Have uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Are pregnant or nursing
* Are unwilling or unable to follow protocol requirements
* Have any condition which in the investigator's opinion deems the subject an unsuitable candidate to participate in this study
* Have metastatic breast cancer
* Have orthopedic or neuromuscular disorders or arthritis that preclude participation in exercise

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2017-10-06 (Actual); Primary Completion 2022-06-02 (Actual); Study Completion 2022-06-02 (Actual)

PRIMARY OUTCOMES:
Proportion of randomized patients who are still on study at the end of the 12 week intervention | At 12 weeks
  The feasibility outcomes will be assessed by a multivariable logistic regression model for the relative odds of remaining on the study (ref: not). Each of the active treatment arms will be compared to the control. The model will be supported by the randomized patient set, counting patients who withdraw from the study as feasibility failures. No variable selection steps will be taken; inferences will be based on the estimates and 95% confidence intervals from the full model. Optimism adjusted odds ratio estimates will also be reported, to better inform design of future studies.

SECONDARY OUTCOMES:
Adherence rate in each of the active intervention arms | Up to 12 weeks
  Will be defined as the proportion of patients on study after 12 weeks who complete ≥ 80% of the intervention activities. One-sided 90% Jeffrey's confidence limits will define a plausible lower limit on the range of values for true (unobserved) feasibility rate for each arm.

OTHER OUTCOMES:
Cardiovascular fitness | At baseline and 12 weeks
  Will determine how it's affected by a 12 week exercise intervention and how it differs by type of intervention program.
Body composition | At baseline and 12 weeks
  Will determine how it's affected by a 12 week exercise intervention and how it differs by type of intervention program.
Quality of life | At baseline and 12 weeks
  Will determine how it's affected by a 12 week exercise intervention and how it differs by type of intervention program. Will be assessed by the Functional Assessment of Cancer Therapy, Breast (FACTB+4).
Cognitive function | At baseline and 12 weeks
  Will determine how it's affected by a 12 week exercise intervention and how it differs by type of intervention program.
Stress and immune function biomarkers | At baseline and 12 weeks
  Will determine how it's affected by a 12 week exercise intervention and how it differs by type of intervention program.
Mitochondrial function | At baseline and 12 weeks
  Will determine how it's affected by a 12 week exercise intervention and how it differs by type of intervention program.

CONTACTS AND LOCATIONS:
Overall Officials: Ellis Levine, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States